CLINICAL TRIAL: NCT00813995
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled, Randomized Study to Evaluate the Safety and Efficacy of the Addition of Sitagliptin 100 mg Once Daily in Patients With Type 2 Diabetes With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: A Study to Test the Safety and Efficacy of Adding Sitagliptin in Patients With Type 2 Diabetes Mellitus (MK0431-074)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-074; 2008_601
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental)
  Interventions: Drug: Comparator: Sitagliptin phosphate
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: Sitagliptin phosphate — All participants will receive placebo tablets two weeks prior to treatment period. Participants will receive sitagliptin phosphate 100 mg tablets once daily (q.d.) and continue on stable dose of metformin therapy (500 or 850 mg twice daily). Treatment period of 24 weeks.
  Other Names: GLUCOPHAGE®
  Arms: Sitagliptin
Drug: Comparator: Placebo — All participants will receive placebo tablets two weeks prior to treatment period. Participants will receive sitagliptin phosphate placebo tablets q.d. and continue on stable dose of metformin therapy (500 or 850 mg twice daily). Treatment period of 24 weeks.
  Other Names: GLUCOPHAGE®
  Arms: Placebo

SUMMARY:
A study to assess the safety and efficacy of the addition of sitagliptin compared to placebo in patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 78 years of age
* Currently on metformin monotherapy

Exclusion Criteria:

* History of Type 1 diabetes mellitus or ketoacidosis
* Currently on a weight loss program and not in the maintenance phase or has started on a weight loss medication within the last 8 weeks
* Has undergone surgery requiring general anesthesia within the past 4 weeks or has planned major surgery
* Currently participating in a study or has participated in a study with or without an investigational compound or device within the past 12 weeks
* History of active liver disease such as chronic active hepatitis B or C, cirrhosis or symptomatic gallbladder disease
* HIV positive
* Pregnant, breast-feeding or planning to become pregnant during the study
* User of recreational or illicit drugs or has a recent history (within the past year) of drug or alcohol abuse or dependence

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2008-12-09 (Actual); Primary Completion 2010-08-09 (Actual); Study Completion 2010-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Yang W, Guan Y, Shentu Y, Li Z, Johnson-Levonas AO, Engel SS, Kaufman KD, Goldstein BJ, Alba M. The addition of sitagliptin to ongoing metformin therapy significantly improves glycemic control in Chinese patients with type 2 diabetes. J Diabetes. 2012 Sep;4(3):227-37. doi: 10.1111/j.1753-0407.2012.00213.x. PMID 22672586

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitagliptin phosphate 100 mg tablets once daily (q.d.) and a stable dose of metformin therapy for 24 weeks.
- Placebo: Placebo tablets q.d. and a stable dose of metformin therapy for 24 weeks.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 197 | 198
Completed | 174 | 182
Not Completed | 23 | 16
Not completed — Clinical adverse event | 9 | 3
Not completed — Laboratory adverse event | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 4 | 2
Not completed — Other reason | 2 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Subject moved | 4 | 0
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 197 | 198 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (9.0) | 55.1 (9.8) | 54.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 90 | 195
  Male | 92 | 108 | 200
Region of Enrollment [Number; unit: participants]
  China | 197 | 198 | 395
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.5 (0.9) | 8.5 (0.9) | 8.5 (0.9)
2-hour Post-meal Glucose [Mean (Standard Deviation); unit: mg/dL] — 392 participants with available data: sitagliptin, n=192; placebo, n=196
  mg/dL | 258.0 (58.0) | 258.7 (63.2) | 258.3 (60.6)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 173.4 (39.3) | 173.9 (40.0) | 173.7 (39.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (defined as a subset of all randomized participants who received at least one dose of double-blind study medication, and had both a baseline [randomization] measurement and a post-randomization measurement) using last observation carried forward for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 191 | 194
Percent | -1.02 (0.99) [-1.16 to -0.87] | -0.14 (1.22) [-0.28 to 0.01]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA — Pairwise comparison

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24 for Participants on Metformin 1000 mg/Day
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Sitagliptin: Sitagliptin phosphate 100 mg tablets once daily (q.d.) and a stable dose of metformin therapy (1000 mg/day) for 24 weeks.
- Placebo: Placebo tablets q.d. and a stable dose of metformin therapy (1000 mg/day) for 24 weeks.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 94 | 97
Percent | -0.84 (1.09) [-1.07 to -0.62] | -0.01 (1.31) [-0.23 to 0.20]

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24 for Participants on Metformin 1700 mg/Day
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Sitagliptin: Sitagliptin phosphate 100 mg tablets once daily (q.d.) and a stable dose of metformin therapy (1700 mg/day) for 24 weeks.
- Placebo: Placebo tablets q.d. and a stable dose of metformin therapy (1700 mg/day) for 24 weeks.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 97 | 97
Percent | -1.14 (0.88) [-1.35 to -0.93] | -0.21 (1.12) [-0.43 to 0.02]

4. Secondary Outcome: Change From Baseline in 2-hour Post-meal Glucose (PMG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 173 | 163
mg/dL | -43.4 (57.3) [-51.5 to -35.3] | -10.0 (60.0) [-18.4 to -1.7]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 191 | 195
mg/dL | -20.3 (39.1) [-26.2 to -14.5] | 0.5 (40.1) [-5.3 to 6.4]

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 7/197 | 5/198
Other Adverse Events (participants affected / at risk) | 10/197 | 13/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=197) | Placebo (N=198)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL CORD INJURY CERVICAL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 2 (2) | 0 (0)
IIIrd NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
EPIGLOTTIC CYST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=197) | Placebo (N=198)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (12) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the multicenter publication or 24 months after study completion, whichever comes first, an investigator may publish the results for their study site independently. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.